CLINICAL TRIAL: NCT06411184
Title: Safety and Efficacy of Treg Cell in the Treatment of GVHD After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Safety and Efficacy of Treg Cell in the Treatment of GVHD
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Kai Lin Xu，MD, professor, Xuzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XYFY2024-KL045-01
Record Dates: First submitted 2024-05-07; First posted 2024-05-13 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: GVHD
Keywords: Regulatory T-Lymphocytes; GVHD

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Regulatory T-Lymphocytes (Experimental): Autologous Regulatory T-Lymphocytes 1*10^6/kg, 2*10^6/kg, 4*10^6/kg and 8*10^6/kg, respectively until restrictive toxic reaction occurs
  Interventions: Drug: Regulator T Cells

INTERVENTIONS:
Drug: Regulator T Cells — Autologous Regulatory T-Lymphocytes 1*10^6/kg, 2*10^6/kg, 4*10^6/kg and 8*10^6/kg, respectively until restrictive toxic reaction occurs
  Other Names: Regulatory T-Lymphocytes

SUMMARY:
This is a randomized, single-center phase 1/2a clinical trial without blinding. Regulatory T cells (Tregs) have shown potential in treating various immune-related diseases, including autoimmune disorders, transplant rejection, and inflammatory diseases. The investigators plan to recruit participants for a clinical trial to evaluate the efficacy and safety of autologous Tregs in the treatment of GVHD.

DETAILED DESCRIPTION:
This randomized, single-center phase 1/2a clinical trial, conducted without blinding, aims to explore the therapeutic promise of regulatory T cells (Tregs). Tregs are specialized immune cells that play a crucial role in modulating the body's immune response, thus offering a unique therapeutic avenue for immune-related conditions. They have already demonstrated significant potential in managing a spectrum of diseases, including autoimmune disorders such as multiple sclerosis and type 1 diabetes, inflammatory conditions like inflammatory bowel disease, and transplant rejection, which is commonly encountered in organ and stem cell transplants. The trial's primary focus is on graft-versus-host disease (GVHD), a severe complication that can occur after allogeneic hematopoietic stem cell transplantation (HSCT). GVHD emerges when the donated immune cells attack the recipient's tissues, leading to symptoms ranging from mild to life-threatening. Currently, GVHD treatment relies on broad immunosuppressive therapies, which often come with significant side effects and may not always be effective. By recruiting participants for this clinical trial, we aim to assess the safety and efficacy of Tregs in mitigating the immune system's attack on the recipient's body. Autologous Tregs offer a more targeted approach due to their ability to distinguish between harmful and beneficial immune responses, potentially reducing the need for broad immunosuppression. The trial's structure includes dose-escalation and dose-expansion phases to evaluate optimal dosages, assess any adverse reactions, and measure the therapeutic benefits in GVHD management. Through this systematic and thorough evaluation, the investigators hope to refine Treg therapy and establish a clear safety profile. Ultimately, this trial seeks to unlock the therapeutic potential of autologous Tregs, paving the way for future applications in a broader range of conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥18 years who have undergone allogeneic hematopoietic stem cell transplantation (allo-HSCT), regardless of gender.
2. Those with persistent manifestations of graft-versus-host disease (GVHD) and suitable for systemic treatment.
3. Previously received at least 1 but not more than 5 lines of systemic treatment for GVHD.
4. Corticosteroid therapy dose stable for the two weeks before screening; or, if taking prednisone or an equivalent dose of other corticosteroids at a dose >0.5mg/kg/day for four weeks, with ongoing GVHD manifestations and no improvement; or, if two attempts to taper steroids to a lower dose have failed, and it is necessary to increase the prednisone dose to >0.25mg/kg/day or an equivalent dose.
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) score: 0~1.
6. Anticipated survival of more than 12 months.

   General criteria:
7. Serum pregnancy test negative for women of childbearing age during the screening period.
8. Sexually active women of childbearing age participating in this study must agree to contraception during the trial and after the last dose of medication.

Exclusion Criteria:

1. Patients who have received experimental treatment for systemic GVHD within the 28 days prior to enrollment, which was effective and could completely alleviate immunosuppression.
2. Blood cancer relapse (according to the corresponding criteria for relapse of the primary blood cancer) or post-transplant lymphoproliferative disease at the time of screening.

   Laboratory tests:
3. Absolute neutrophil count (ANC) <1.5×10^9/L (excluding GVHD as the cause).
4. Platelet count <50×10^9/L (excluding GVHD as the cause).
5. Alanine aminotransferase (ALT) >3 times the upper limit of normal (ULN), aspartate aminotransferase (AST) >3×ULN (excluding GVHD as the cause).
6. Total bilirubin (TBIL) >1.5×ULN (excluding GVHD as the cause).
7. Creatinine clearance CrCl <60 mL/min (Cockcroft-Gault formula).

   General criteria:
8. Pregnant or lactating women.
9. History of serious illness or other evidence indicating a serious illness, or any other condition that the investigator believes may make the subject unsuitable for this study.

   * History of severe cardiovascular disease [New York Heart Association (NYHA) functional class III or IV], including but not limited to ventricular arrhythmias requiring clinical intervention, uncontrolled hypertension (systolic blood pressure ≥160mmHg and/ or diastolic blood pressure ≥100mmHg); within 6 months prior to enrollment, there is unstable angina, acute coronary syndrome, congestive heart failure, stroke, or other cardiovascular events of class III or above; at screening, NYHA functional class ≥II or left ventricular ejection fraction (LVEF) <50% on echocardiography.
   * Unable to take oral medications, with severe (NCI CTCAE v5.0 ≥ grade 3) chronic gastrointestinal dysfunction, the presence of malabsorption syndrome, or any other condition affecting gastrointestinal absorption.
   * History of clear neurological or psychiatric disorders (including epilepsy or dementia), currently suffering from psychiatric disorders, or judged by the investigator to be non-compliant and unsuitable for participation in the study.
   * History of other severe (NCI CTCAE v5.0 ≥ grade 3) systemic diseases, deemed unsuitable for participation in the clinical trial by the investigator.
10. Other circumstances in which the investigator deems it inappropriate to participate in this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Baseline up to 60 days after taking Iguratimod]
  Adverse events assessed according to NCI-CTCAE v5.0

SECONDARY OUTCOMES:
complete response (CR) | Month 1, 2, 3 and 4
  Assessment of CR at Month 1, 2, 3 and 4. According to the CHRONIC GVHD ACTIVITY ASSESSMENT - CLINICIAN recorded in NIH Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease: IV. The 2014 Response Criteria Working Group report. (Biol Blood Marrow Transplant. 2015 Jun;21(6):984-99.)
partial response (PR) | Month 1, 2, 3 and 4
  Assessment of CR at Month 1, 2, 3 and 4. According to the CHRONIC GVHD ACTIVITY ASSESSMENT - CLINICIAN recorded in NIH Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease: IV. The 2014 Response Criteria Working Group report. (Biol Blood Marrow Transplant. 2015 Jun;21(6):984-99.)
stable disease (SD) | Month 1, 2, 3 and 4
  Assessment of CR at Month 1, 2, 3 and 4. According to the CHRONIC GVHD ACTIVITY ASSESSMENT - CLINICIAN recorded in NIH Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease: IV. The 2014 Response Criteria Working Group report. (Biol Blood Marrow Transplant. 2015 Jun;21(6):984-99.)
progressed disease (PD) | Month 1, 2, 3 and 4
  Assessment of CR at Month 1, 2, 3 and 4. According to the CHRONIC GVHD ACTIVITY ASSESSMENT - CLINICIAN recorded in NIH Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease: IV. The 2014 Response Criteria Working Group report. (Biol Blood Marrow Transplant. 2015 Jun;21(6):984-99.)